CLINICAL TRIAL: NCT05641519
Title: Skills-Based Educational Strategies for Reduction of Vascular Events in Orange County
Acronym: SERVEOC
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, Irvine (Other)
Collaborators: National Institutes of Health (NIH) (NIH); Ohio State University (Other); Latino Health Access (Unknown); Vietnamese American Cancer Foundation (Unknown); Radiate Consulting (Unknown); National Institute on Minority Health and Health Disparities (NIMHD) (NIH)
Responsible Party: Principal Investigator, Bernadette Boden-Albala, Director and Founding Dean, University of California Irvine Program in Public Health, Professor, Departments of Health, Society and Behavior (Program in Public Health) and Neurology (School of Medicine), Susan and Henry Samueli College of Health Sciences, University of California, Irvine
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 283; 5P50MD017366-04 (NIH)
Record Dates: First submitted 2022-09-16; First posted 2022-12-07 (Actual); Last update posted 2025-09-09 (Actual); Status verified 2025-05

CONDITIONS: Hypertension
Keywords: Hypertension; Life's Essential 8; Social Networks; Community Health Workers; Hispanic/Latinx; Vietnamese
MeSH Terms: conditions — Hypertension | interventions — Standard of Care

STUDY DESIGN:
Intervention Model Description: SERVE OC is a randomized controlled trial that utilizes block randomization, and the family/household will be the unit of randomization (participants in the same household will be randomized to the same intervention arm). We will prospectively enroll 150-200 households with school-age children from the SAC cohort and randomize the Hispanic/Latinx, Vietnamese, and non-Hispanic/ Vietnamese households to the SERVE OC intervention or enhanced standard intervention (ESI) to ensure balance between intervention arms within each race and ethnic group. Participant follow-up will occur at 12, 24, and 36 months.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Enhanced Standard Intervention (Placebo Comparator): Families randomized to enhanced standard intervention (ESI) will be given informational materials from the American Heart Association on cardiovascular health. ESI includes self-management which is standard care. At 12, 24, and 36 months they will be asked to return for in person follow-up to collect bio measures again and complete follow up surveys at the UCI FQHC in Santa Ana or during scheduled community data collection events. All adults will be asked to take their blood pressure with the device once a week.
  Interventions: Behavioral: Enhanced Standard Intervention
- SERVE OC Intervention (Experimental): In the SERVE OC intervention, participants will receive AHA informational materials, access to the app/web portal, and will be assigned a CHW to work with over the 3 years of the study. The CHW will facilitate the intervention for the family which includes 1) Conducting a family "intake" of risk factors through the LE8 assessment 2) Facilitate the creation of a family network-tailored action plan 3) Provide guidance to activate/reinforce action plans using the interactive part of the app/web portal. They will meet with their CHW monthly to learn about CVH, work on their goals, and action plans. Meetings with CHWs will take place in their homes, the UCI FQHC in Santa Ana, over zoom, or other locations. All adults will be asked to take their blood pressure with the device once a week.
  Interventions: Behavioral: SERVE OC Intervention

INTERVENTIONS:
Behavioral: SERVE OC Intervention — SERVE OC intervention for the family which includes 1) Conducting a family "intake" of risk factors through the LE8 assessment and discussing prevention/risk reduction 2) Facilitate the creation of a family network-tailored action plan 3) Provide guidance to activate/reinforce action plans using the interactive part of the app/web portal. They will meet with their CHW monthly to learn about CVH, work on their goals, and action plans. Meetings with CHWs will take place in their homes, the UCI FQHC in Santa Ana, over zoom, or other locations such as local churches, parks, community centers, or grocery stores (for field trips) They will also receive messages from them throughout the duration of the study using their preferred method of contact (text, email, webportal/app, phone call) for reinforcement and scheduling meetings
  Other Names: Community Health Worker Intervention; Family Based Intervention
  Arms: SERVE OC Intervention
Behavioral: Enhanced Standard Intervention — Enhanced Standard Intervention will be given informational materials from the American Heart Association on cardiovascular health. ESI includes self-management which is standard care
  Other Names: Usual Care; Standard of Care
  Arms: Enhanced Standard Intervention

SUMMARY:
The Skills-Based Educational strategies for Reduction of Vascular Events in Orange County, CA (SERVE OC) study aims to evaluate the efficacy of a culturally tailored, skills-based, cardiovascular health (CVH) intervention amongst a cohort of Latinx and Vietnamese families in Santa Ana, CA. The SERVE OC intervention was adapted from our previous work, the Discharge Educational Strategies for Reduction of Vascular Events (DESERVE) intervention, for the primordial prevention of hypertension (HTN) and other risk factors for cardiovascular disease (CVD). (The DESERVE study was conducted at New York University under their IRB). The intervention will be delivered by community health workers (CHWs) and will focus on: 1) optimizing risk perception, 2) enhancing provider-family communication, and 3) identifying challenges to CVH. Participants will receive multi-lingual materials and access to an app/web portal to identify healthy goals and strategies around modifiable risk factors for CVH, Life's Essential 8. SERVE OC will follow participants for 36-months to examine changes in CVH using Life's Simple 7 (LS7): smoking status, physical activity, weight, diet, blood glucose, cholesterol, and blood pressure (BP) scores and changes in systolic blood pressure (SBP) among adult participants versus enhanced standard intervention (ESI). Remote blood pressure (BP) monitoring will also be used to assess BP over time. CHWs will engage families in identifying barriers to CVH and solutions to share with community stakeholders. Using this community-based research (CBPR) approach the investigators hope to improve health equity within the community through enhanced social capital, empowerment, and advocacy capacity. This study is part of a multi-center projected coordinated by the UCLA-UCI Center for Eliminating Cardio-Metabolic Disparities in Multi-Ethnic Populations (UC END-DISPARITIES), aimed at improving CVH among underserved populations in Los Angeles and Orange County.

DETAILED DESCRIPTION:
1. Participants from the Santa Ana Cares (SAC) cohort will be invited to participate in SERVE OC until projected sample size is reached. Vietnamese households will be over sampled to enhance recruitment of this population.
2. Informed consent/parent permission/assent will be collected from eligible participants who agree to participate in the study. The study team and trained CHWs, will collect informed consent.
3. Families will then be randomized into SERVE OC or to Enhanced Standard Intervention (ESI)
4. The study team, will conduct baseline assessments for each family. Baseline assessments includes a bio-measure assessment which includes measuring blood pressure, height, weight, waist circumference, HbA1c, and cholesterol. During baseline, participants will also answer questions about diet, physical activity, sleep, their vascular health, socio-demographics, and behavioral, social network, and health equity measures. The CHWs will be trained and will help the study team with administering the participant surveys. CHWs will be UCI affiliated and all CHWs will be added to the research personnel tracking log. All study team members will also be added to the research personnel tracking log.
5. Families randomized to ESI will be given informational materials from the American Heart Association on cardiovascular health. ESI includes self-management which is standard care. At 12, 24, and 36 months they will be asked to return for in person follow-up to collect bio measures again and complete follow up surveys during scheduled community data collection events.
6. Families randomized to SERVE OC will receive AHA informational materials, access to the app/web portal, and will be assigned a CHW to work with over the 3 years of the study. The CHW will facilitate the SERVE OC intervention for the family which includes 1) Conducting a family "intake" of risk factors through the LE8 assessment and discussing prevention/risk reduction 2) Facilitate the creation of a family network-tailored action plan 3) Provide guidance to activate/reinforce action plans using the interactive part of the app/web portal. They will meet with their CHW monthly to learn about CVH, work on their goals, and action plans. Meetings with CHWs will take place in their homes, the UCI FQHC in Santa Ana, over zoom, or other locations such as local churches, parks, community centers, or grocery stores (for field trips) They will also receive messages from them throughout the duration of the study using their preferred method of contact (text, email, web portal/app, phone call) for reinforcement and scheduling meetings. Families will be asked to return for follow-up at 12, 24, and 36 months to collect bio measures and complete follow up surveys/interviews.

   a. CHWs: CHWs will be UCI affiliated. All CHWs will be added to the research personnel tracking log. Over the 3 years of the study, the CHWs will interact with families in their home, or at community sites depending on the family's preference. They will encourage family level activities to improve CVH using interactive curriculums, narrative videos, informational workbooks (available in Spanish, Vietnamese, or English), the web portal/app, and reinforcement. They will ask families to identify barriers to improving CVH and possible solutions to utilize later for SERVE OC community activities. CHWs will also respond to other issues families may have including poverty, food insecurity, domestic abuse, and substance misuse. After 1 year, the team will incorporate relevant educational materials and protocols into the intervention to help CHWs respond to these issues and to provide families with resources.

   App/Web portal: For SERVE OC, the existing FURRThERhealth.com interactive web portal/app which was used in previous studies will be updated for the needs of the SERVE OC intervention. The web portal will facilitate the creation of tailored action plans, including setting goals and planning activities; allow groups to track activities and earn stars and trophies for their accomplishments; facilitate online communication in preferred languages; and provides curated AHA and other resources to support primary and secondary prevention. During the initial meeting, the CHW will introduce the portal to families. Each individual will be assigned a unique profile with corresponding avatar handle that is linked to their identifying information. With the CHW, the login process and site functionality will be demonstrated to all members of the group. Tech support information will be made available. There are 2 sections of the web portal: 1) the resource section and 2) the facilitated network engagement (goal creation, activity tracking, chat and photo sharing, push notifications and e-messages). The CHW will work with the families to enter chosen goals and activities into the portal and demonstrate the process of tracking activity completion. After goal setting, families will start to receive push messages about working together on healthy lifestyle and risk reduction. The initial messages focus on support for the transition to engaging in healthy lifestyles as a family. The investigators anticipate that there will be changes to goals and times when networks go into holding patterns (no activity or motivation). Messages from SERVE OC will change to address new barriers and challenges.
7. All participants will also be invited to attend community events, which will occur a few time a year. At these events the study team will facilitate discussions between community members, community health organizations, local government, and subject matter experts to identify issues and possible solutions to improve health the community of Santa Ana. Food, childcare, and fun, healthy, educational activities will be provided for all.
8. All families/household will receive a Withings BPM Connect, which is a remote blood pressure measuring monitor, that allows their blood pressure readings to be sent directly to our research team through an online cloud to allow us to examine BP trends over time. All participating adult family members, 18 years of age and older, will be asked to take their blood pressure readings once a week. The study team will teach them how to use the blood pressure monitor and provide them with instructions to take home. If they are in the SERVE OC intervention the CHWs will ask them how they are doing with the weekly BP readings or remind them to take their measurements using the app/web portal.
9. The investigators will also conduct focus groups throughout the 3 years of the study as the SERVE OC intervention is iterative and will be informed by community stakeholders as it goes on. This is a CBPR practice.
10. At baseline and 3 years, COVID-19 antibody testing will be conducted.

ELIGIBILITY:
Inclusion Criteria:

1. Living in Santa Ana, Anaheim, Westminster or Garden Grove
2. Speaks one of the languages in which the survey is administered in (English, Spanish, and Vietnamese)
3. Aged >=18 years old at time of enrollment
4. Has at least one friend/family/household member participating in the study with them, (if they are a minor they must have at least one adult participant participating with them)
5. If child turns 5 during the 3 years of the study they will be eligible to participate and we will enroll them with parent permission

Exclusion Criteria:

1. Dementia history, cognitive impairment, or any condition impairing his/her ability to participate in education
2. Life expectancy less than 1 year
3. Unable to give informed consent or unable to obtain parent/guardian permission (minors)
4. Lives in a nursing home or requires 24-hour care

Min Age: 5 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 483 (Actual)
Dates: Start 2022-11-18 (Actual); Primary Completion 2026-07 (Estimated); Study Completion 2026-07 (Estimated)

PRIMARY OUTCOMES:
Life's Essential 8 | Baseline
  To evaluate the efficacy of family-based SERVE OC intervention versus ESI in achieving ""ideal" cardiovascular health as measured by Life's Essential 8 (LE8). LE8 is an assessment composed of 8 domains: smoking status, physical activity, weight, diet, sleep, blood glucose, cholesterol, and blood pressure (BP). LE8 scores can be calculated using the My Life Check portal from the American Heart Association. Having four or more ideal LE8 domains out of the total 8 domains will be considered 'ideal CVH'. The outcome is the number of LE8 domains that are ideal out of the total 8 domains.
Life's Essential 8 | 1 year
  To evaluate the efficacy of family-based SERVE OC intervention versus ESI in achieving ""ideal" cardiovascular health as measured by Life's Essential 8 (LE8). LE8 is an assessment composed of 8 domains: smoking status, physical activity, weight, diet, sleep, blood glucose, cholesterol, and blood pressure (BP). LE8 scores can be calculated using the My Life Check portal from the American Heart Association. Having four or more ideal LE8 domains out of the total 8 domains will be considered 'ideal CVH'. The outcome is the number of LE8 domains that are ideal out of the total 8 domains.
Life's Essential 8 | 2 year
  To evaluate the efficacy of family-based SERVE OC intervention versus ESI in achieving ""ideal" cardiovascular health as measured by Life's Essential 8 (LE8). LE8 is an assessment composed of 8 domains: smoking status, physical activity, weight, diet, sleep, blood glucose, cholesterol, and blood pressure (BP). LE8 scores can be calculated using the My Life Check portal from the American Heart Association. Having four or more ideal LE8 domains out of the total 8 domains will be considered 'ideal CVH'. The outcome is the number of LE8 domains that are ideal out of the total 8 domains.
Life's Essential 8 | 3 year
  To evaluate the efficacy of family-based SERVE OC intervention versus ESI in achieving ""ideal" cardiovascular health as measured by Life's Essential 8 (LE8). LE8 is an assessment composed of 8 domains: smoking status, physical activity, weight, diet, sleep, blood glucose, cholesterol, and blood pressure (BP). LE8 scores can be calculated using the My Life Check portal from the American Heart Association. Having four or more ideal LE8 domains out of the total 8 domains will be considered 'ideal CVH'. The outcome is the number of LE8 domains that are ideal out of the total 8 domains.

SECONDARY OUTCOMES:
Systolic Blood Pressure | Baseline
  To examine the effect of SERVE OC intervention versus ESI in changing systolic blood pressure (SBP) among adults.
Systolic Blood Pressure | Year 1
  To examine the effect of SERVE OC intervention versus ESI in changing systolic blood pressure (SBP) among adults.
Systolic Blood Pressure | Year 2
  To examine the effect of SERVE OC intervention versus ESI in changing systolic blood pressure (SBP) among adults.
Systolic Blood Pressure | Year 3
  To examine the effect of SERVE OC intervention versus ESI in changing systolic blood pressure (SBP) among adults.

CONTACTS AND LOCATIONS:
Overall Officials: Bernadette Boden-Albala, DrPH, MPH, Principal Investigator — UCI Program in Pubic Health
Locations (1):
- University of California, Irvine, Irvine, California, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Boden-Albala B, Draughter-Espinoza D, Castro M, Gutierrez D, Cardenas C, Landry MJ, Wing J, Albala B. Knowledge, barriers, and facilitators for promoting cardiovascular health in a Latino community: a qualitative sub-study of the Skills-based Educational Strategies for Reduction of Vascular Events in Orange County. Front Public Health. 2025 Jun 18;13:1531775. doi: 10.3389/fpubh.2025.1531775. eCollection 2025. PMID 40606080